CLINICAL TRIAL: NCT04189120
Title: Evaluation the Effect of Ultrasound Guided Superficial, Deep Serratus Plane Blocks and Thoracic Epidural in Cancer Patients Undergoing Thoracotomy: A Prospective Randomized Controlled Study
Brief Title: The Effect of Ultrasound Guided Superficial, Deep Serratus Plane Blocks and Thoracic Epidural in Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AP1811-30102
Record Dates: First submitted 2019-04-22; First posted 2019-12-06 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Post-thoracotomy Pain Syndrome
Keywords: post thoracotomy pain; thoracic epidural; serratus anterior plane block; ultrasound
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic epidural analgesia (TEA) (Active Comparator): Under full aseptic conditions and wearing sterile gloves while the patient is in setting position, skin infiltration will be done with 2 ml of 1% lidocaine, then an 18-G Epidural needle with a 20-G catheter (Perifix, B.Braun, Germany) will be inserted through the T6-T7 interspace, and the epidural space located using the loss of resistance technique. The catheter then advanced approximately 3 cm cephalic. A test dose of 3 ml of 1% lidocaine containing epinephrine in a ratio of 1:200,000 administered to detect unintentional intrathecal or IV injection. After negative response, 15 ml of 0.25% epidural bupivacaine will be injected and the patient will be turned to the supine position.
  Interventions: Procedure: Thoracic epidural analgesia , superficial serratus plane block and deep serratus plane block
- Ultrasound-guided superficial serratus plane block (SSPB) (Active Comparator): Under full aseptic conditions, the patient is placed in lateral position with the diseased side up, sterile field is established with a povidone iodine solution, and the linear transducer 8-12 MH (sonosite M-turbo ; Inc., Bothell, WA, USA) is covered by a disposable sterile cover and will be placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The ribs will be counted until the fifth rib is identified in the mid-axillary line. The muscles will be identified easily overlying the fifth rib, the latissimus dorsi , teres major and serratus muscles . A skin wheal of 1% lidocaine will be made 1 cm away from the lateral edge of the transducer thorough which the needle (22-G, 50-mm Touhy needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle beneath the latissimus dorsi. Under continuous ultrasound guidance 30 ml of 0.25% bupivacaine will be injected
  Interventions: Procedure: Thoracic epidural analgesia , superficial serratus plane block and deep serratus plane block
- Ultrasound-guided deep serratus plane block (DSPB) (Active Comparator): Under full aseptic conditions, the patient is placed in lateral position with the diseased side up, sterile field is established with a povidone iodine solution, and the linear transducer 8-12 MH (sonosite M-turbo ; Inc., Bothell, WA, USA) is covered by a disposable sterile cover and will be placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The ribs will be counted until the fifth rib is identified in the mid-axillary line. A skin wheal of 1% lidocaine will be made 1 cm away from the lateral edge of the transducer thorough which the needle (22-G, 50-mm Touhy needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane between the posterior border of the serratus anterior muscle and the corresponding surface of the rib. Under continuous ultrasound guidance 30 ml of 0.25% bupivacaine will be injected deep to the serratus muscle separating the serratus anterior muscle from the external intercostal muscle.
  Interventions: Procedure: Thoracic epidural analgesia , superficial serratus plane block and deep serratus plane block

INTERVENTIONS:
Procedure: Thoracic epidural analgesia , superficial serratus plane block and deep serratus plane block — neuroaxial thoracic epidural analgesia and regional analgesia supeficial and deep serratus plane blocks

SUMMARY:
Pain after thoracotomy is known to be sever acute pain that is resulted from retraction, resection or fracture of ribs .This pain increases post operative morbidity and if not properly managed peri-operatively, chronic post thoracotomy pain syndrome may develop. Different methods are described to manage post thoracotomy pain.Thoracic epidural analgesia is believed to be the corner stone in the peri-operative care for thoracotomy providing the most effective analgesia. Serratus anterior plane (SAP) block has recently been described as a regional anesthetic technique to provide analgesia for thoracic wall surgeries. During SAP block, local anesthesia are deposited in the fascial plane either superficial to the serratus muscle or deep to the serratus anterior muscle in the mid-axillary line . Serratus anterior block provides analgesia to a hemithorax by blocking the lateral branches of the intercostal nerves. This study aims To compare the effect of superficial, deep serratus plane blocks and thoracic epidural analgesia in maintaining hemodynamic and controlling post thoracotomy pain.

DETAILED DESCRIPTION:
The aim of thoracotomy surgery is to explore the thoracic cavity and manage different pathologies including pulmonary, diaphragmatic, mediastinal, esophageal and vascular pathologies. It can be performed posterolaterally, anterolaterally or even anteriorly.

Pain after thoracotomy is known to be sever acute pain that is resulted from retraction, resection or fracture of ribs and dislocation of costovertebral joints; injury of intercostal nerves or even irritation of the pleura by chest tubes inserted at the end of surgery. This pain increases post-operative morbidity and if not properly managed peri-operatively, chronic post thoracotomy pain syndrome may develop.

Different methods are described to manage post thoracotomy pain. Intravenous (IV) drugs such as opioids and non-steroidal anti-inflammatory drugs (NSAIDS), infiltration of local anesthetics to the wound and regional anesthetic techniques such as thoracic epidural analgesia (TEA), paravertebral block, intercostal block and intra/extra pleural block are methods frequently used to relieve post thoracotomy pain.

Thoracic epidural analgesia is believed to be the corner stone in the peri-operative care for thoracotomy providing the most effective analgesia. However, thoracic epidural analgesia is associated with serious complications such as hypotension, dural puncture with the needle or the catheter, post-dural puncture headache, respiratory depression with adding opioids, spinal cord injury and anterior spinal artery syndrome.

The serratus muscle is a superﬁcial and easily identified muscle that is considered a true landmark to implement thoracic wall blocks because the intercostal nerves pierce it.Serratus anterior plane (SAP) block has recently been described as a regional anesthetic technique to provide analgesia for breast and thoracic wall surgeries. During SAP block, local anesthesia are deposited in the fascial plane either superficial to the serratus muscle or deep to the serratus anterior muscle in the mid-axillary line .Serratus anterior block provides analgesia to a hemithorax by blocking the lateral branches of the intercostal nerves.SAP block is also expected to avoid autonomic blockade associated with TEA and other complications involving the pleura and central neuraxial structures.

Ultrasound imaging made the practice of regional anesthesia easier in visualization and identification of usual and unusual position of nerves , blood vessels , needle during its passage through the tissues, as well as deposition and spread of local anesthetics in the desired plane and around the desired nerve.

ELIGIBILITY:
Inclusion Criteria:

1. ASA(American Society of Anesthesia) class I and II.
2. Age ≥ 18 and ≤ 60 Years.
3. Patients undergoing thoracic surgery eg: lobectomy, pneumonectomy or pleuro-pneumonectomy

Exclusion Criteria:

1. Patient refusal.
2. Local infection at the puncture site.
3. Coagulopathy with INR ( international normalized ratio ) ≥ 1.6: hereditary (e.g. hemophilia, fibrinogen abnormalities & deficiency of factor II) - acquired (e.g. impaired liver functions with prothrombin concentration less than 60 %, vitamin K deficiency & therapeutic anticoagulants drugs).
4. Unstable cardiovascular disease.
5. History of psychiatric and cognitive disorders.
6. Patients allergic to medication used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
changes and stability of Mean Arterial Blood Pressure (MAP). | every 5 minutes for 3 hours during the surgey
  Mean arterial blood pressure to be measured after completion of intervention in patients with thoracotomies then every five minutes till the end of surgery.

SECONDARY OUTCOMES:
Total intra-operative fentanyl consumption | 2-3 hours (Surgery time) surgery
  the rescue analgesia will be administered intra-operative by fentanyl IV and the total fentanyl used will be recorded and compared between the groups
Pain scores using Visual analogue score | 24 hours after the surgery
  Pain scores using Visual analogue score (VAS) (0 mm = no pain to 10mm = worst pain imaginable) at predetermined time intervals (1, 2, 6, 12 and 24h) postoperative.
1st time opioids requested post-operative. | 24 hours after the surgery
  In case of postoperative pain recorded, rescue analgesia will be provided as IV morphine (3 mg) then continuous infusion of morphine through Patient Controlled Analgesia ( PCA ) to keep the VAS scores<3. The total 24-hour morphine consumption will be recorded for every patient.
Total morphine consumption. | 24 hours after the surgery
  The total 24-hour morphine consumption will be recorded for every patient post operative.

CONTACTS AND LOCATIONS:
Overall Officials: Ekramy Mansour, MD, Study Director — National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989